CLINICAL TRIAL: NCT05263427
Title: Maternal-Fetal Monitoring by Connected Abdominal Patch - MOMA
Acronym: MOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); BioSerenity (Industry); National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021_0548; 2022-A00107-36 (Other: ID-RCB number, ANSM); ANR-18-CE19-0015-01 (Other: AAP number, ANR)
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Obstetrical Complications; Monitoring Injury of Scalp of Newborn
Keywords: Fetal Heart Rate; Monitoring; Uterine contraction; Electrocardiogram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOCONAUTE and gold standard : cardiotocograph (Experimental)
  Interventions: Device: TOCONAUTE

INTERVENTIONS:
Device: TOCONAUTE — This study will be carried out during delivery. The will be placed on the mother's abdomen to capture fetal and maternal heart rate as well as the uterine contractions in parallel of the cardiotocograph.
  For each of the participants, the TOCONAUTE will remain on the mother's abdomen till childbirth. This procedure will not affect the usual care of the patient.
  Other Names: foetal heart rate and uterine contractions recording

SUMMARY:
During a previous clinical trial (RCF-abdo: 2018-A01194-51), trans-abdominal signals were collected in 90 patients at the maternity Jeanne de Flandre. This database allowed us to develop a new medical device able to measure in real time and continuously the fetal heart rate and the uterine contractions.

The goal here is to assess the performance of the device in real situation during labour.

This study will be carried out in the maternity labor ward in CHU Lille, France.

The TOCONAUTE will be placed on the mother's abdomen to capture fetal and maternal heart rate as well as the uterine contractions in parallel of the cardiotocograph.

For each of the participants, the TOCONAUTE will remain on the mother's abdomen till childbirth. This procedure will not affect the usual care of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman in labor
* Singleton
* Cephalic presentation

Exclusion Criteria:

* Hospitalisation for a medical termination of pregnancy
* Death in utero
* Multiple pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — PRegnant women
Enrollment: 60 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Fetal heart rate with the TOCONAUTE | 1 year
  The fetal heart rate from the our device will be averaged on 3 beats and resampled at 4Hz to be comparable to the fetal heart rate from the cardiotocograph.
  Both of the signals will be resynchronized and compared sample by sample with a Pearson's correlation test.
  Measure of the fetal heart rate with the TOCONAUTE compared to the measure of the fetal heart rate with a cardiotocograph.

SECONDARY OUTCOMES:
Uterine contractions with the TOCONAUTE according to the different phase of labor. | 1 year
  Measure of the uterine contractions with the TOCONAUTE compared to the measure of the uterine contractions with a cardiotocograph according to the different phase of labor.
  Both signals of the uterine contractions will be resynchronized and compared sample by sample with a Pearson's correlation test.
Maternal heart rate with the TOCONAUTE | 1 year
  Measure of the maternal heart rate with the TOCONAUTE compared to the measure of the maternal heart rate with a cardiotocograph.
  Both signals of the maternal heart rate will be resynchronized and compared sample by sample with a Pearson's correlation test.
Fetal heart rate with the TOCONAUTE according to the different phase of labor. | 1 year
  Measure of the fetal heart rate with the TOCONAUTE compared to the measure of the fetal heart rate with a cardiotocograph according to the different phase of labor.
Fetal stress index (Heart rate variability index reflecting parasympathetic fluctuation) | 1 year
  Feasibility of the measure of the Fetal stress index (Heart rate variability index reflecting parasympathetic fluctuation)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Garabedian, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France

REFERENCES:
- [Result] Wojtanowski A, Garabedian C, Charlier P, Prot P, Ghesquiere L, De Jonckheere J. Intrapartum monitoring of the fetal heart rate using transabdominal electrocardiography: A reliability and accuracy study. J Gynecol Obstet Hum Reprod. 2025 May;54(5):102942. doi: 10.1016/j.jogoh.2025.102942. Epub 2025 Mar 16. PMID 40101837